CLINICAL TRIAL: NCT04800770
Title: Phosphate Levels of COVID-19 Patients and Mortality
Brief Title: The Effect of COVID-19 Patients' Serum Phosphate Level on Mortality in ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, medical doctor, Ankara City Hospital Bilkent
Other Study IDs: E1-21-1584
Record Dates: First submitted 2021-03-10; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Phosphate Deficiency; Covid19; Mortality
Keywords: COVID19; phosphate deficiency; 4C mortality score
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 4C mortality score — 4C mortality score and phosphate levels

SUMMARY:
The investigators aimed to investigate the relationship between phosphate level and mortality using the 4C Mortality Score in COVID-19 patients who were followed up in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Participants hospitalized in the intensive care unit diagnosed with COVID-19 will incluse in the study

Exclusion Criteria:

* there is no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants hospitalized in the intensive care unit diagnosed with COVID-19 will incluse in the study
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
4C mortality score | 6 months
  4C Mortality Scores of the patients will be calculated, according to age, gender, number of comorbidities, respiratory rate, SpO2, GCS, urea, and CRP parameters
serum phosphate levels | 6 months
  mg/dl
mortality | 28 days
  mortality percentage of patients in 28 days

CONTACTS AND LOCATIONS:
Overall Officials: betül aytaç, MD, Principal Investigator — ankara ch bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Murer H, Forster I, Biber J. The sodium phosphate cotransporter family SLC34. Pflugers Arch. 2004 Feb;447(5):763-7. doi: 10.1007/s00424-003-1072-5. Epub 2003 May 16. PMID 12750889
- [Result] Pistolesi V, Zeppilli L, Polistena F, Sacco MI, Pierucci A, Tritapepe L, Regolisti G, Fiaccadori E, Morabito S. Preventing Continuous Renal Replacement Therapy-Induced Hypophosphatemia: An Extended Clinical Experience with a Phosphate-Containing Solution in the Setting of Regional Citrate Anticoagulation. Blood Purif. 2017;44(1):8-15. doi: 10.1159/000453443. Epub 2017 Feb 21. PMID 28219057
- [Result] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570